CLINICAL TRIAL: NCT04303468
Title: The Effects of a GABA Supplement Versus a Placebo on Glucose Tolerance and Blood Pressure in Prediabetics
Brief Title: Intervention With a GABA Supplement in Prediabetics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: Nunhems (Unknown); Agrico Research (Unknown); Avebe (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NL73194.081.20
Record Dates: First submitted 2020-03-04; First posted 2020-03-11 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Prediabetes; Hypertension
MeSH Terms: conditions — Prediabetic State; Hypertension | interventions — gamma-Aminobutyric Acid

STUDY DESIGN:
Intervention Model Description: Randomized placebo controlled double blind parallel study design
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GABA (Experimental): GABA is a nutrient commonly present in our diet in for example tomatoes and potatoes. It is also commercially sold as dietary supplement. A dose of 500 mg, 3 times daily is used
  Interventions: Dietary Supplement: GABA
- Placebo (Placebo Comparator): The placebo consists of capsules containing powdered cellulose.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: GABA — The dietary supplement GABA will be taken orally 3 times daily, before each main meal
  Arms: GABA
Other: Placebo — Gelatin capsule containing powdered cellulose
  Arms: Placebo

SUMMARY:
In this double-blind parallel placebo controlled intervention study the effects of 3 times daily 500 mg gamma-aminobutyric acid (GABA) supplementation on glucose tolerance and cardiovascular health will be assessed in prediabetics.

ELIGIBILITY:
Inclusion Criteria:

* Age between 50 and 70
* BMI higher or equal to 27 kg/m2
* Impaired fasting glucose (fasting glucose ≥ 6.1 and ≤ 6.9 mmol/L) or/and
* Impaired glucose tolerance (glucose levels ≥ 7.8 and ≤ 11.1 mmol/L, 2-hours after an OGTT or/and glucose levels ≥8.6 mmol/L, 1-hour after an OGTT)

Exclusion Criteria:

* Has been diagnosed with diabetes
* Having other conditions, like liver, pancreatic, cardiovascular, gastro-intestinal or endocrine diseases, that could influence the study results
* Use of medications or supplements that could influence the study results
* Sensitive to medical skin adhesives
* More than 5kg weight change in the past 12 weeks
* Excessive alcohol consumption (>21 glasses/week for men and >14 glasses/week for women on average)
* Being an employee of Wageningen University, division Human Nutrition and Health
* Currently a research subject in other research

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2020-09-29 (Actual); Primary Completion 2021-09-08 (Actual); Study Completion 2021-09-08 (Actual)

PRIMARY OUTCOMES:
Postprandial glycaemic response during a 2 hour oral glucose tolerance test (OGTT) | blood will be drawn at baseline and after 30, 60 and 120 minutes, before and after the 12 weeks intervention
  A 2 hour oral glucose tolerance test with 75gr glucose

SECONDARY OUTCOMES:
Postprandial insulin and glucagon response during a 2 hour OGTT, | blood will be drawn at baseline and after 30, 60 and 120 minutes, before and after the 12 weeks intervention
  A 2 hour oral glucose tolerance test with 75gr glucose
Plasma free fatty acids | before and after the 12 weeks intervention
HbA1c | before and after the 12 weeks intervention
Glucose variability | 5 days during which they eat their habitual diet, before and after the 12 weeks intervention
  The participants wear a flash glucose monitoring sensor with which their interstitial glucose is measured every 15 minutes.
Blood pressure | Dynamic measurement: 24 hours, before and after the 12 weeks intervention
  Single measurement and a dynamic measurement:
  * Mean day systolic and diastolic blood pressure
  * Mean night systolic and diastolic blood pressure
  * Time below or above 120/80 mmHg
Heart rate | before and after the 12 weeks intervention
Concentrion of markers of inflammation in blood | before and after the 12 weeks intervention
  C-reactive protein and cytokines like IL-6 and TNF-alpha
Concentration of triglycerides in blood | before and after the 12 weeks intervention
Concentration of LDL and HDL cholesterol in blood | before and after the 12 weeks intervention
Concentration of ALAT and ASAT in blood | before and after the 12 weeks intervention
Acute effects of GABA on postprandial glucose | 2 hours, after a single administration of 500 mg GABA
  Assessed with an OGTT during which interstitial glucose is measured with flash glucose monitoring
Acute effects of GABA on blood pressure | for 24 hours during which GABA is taken 3 times, each time before the main meal
  Assessed with an ambulatory blood pressure monitor
Sleep quality | before and after the 12 weeks intervention
  Pittsburgh Sleep Quality Index (PSQI) questionnaire, the outcome is a global PSQI score (range: 0-21), with higher scores indicating poorer sleep quality.
Feelings of depression | before and after the 12 weeks intervention
  Patient Health Questionnaire (PHQ-9), the higher the score the more depressed a person is.
Feelings of anxiety | before and after the 12 weeks intervention
  General Anxiety Disorder (GAD-7) questionnaire, the higher the score, the more anxious a person is.
Plasma GABA concentration | before and after the 12 weeks intervention
Plasma glutamate concentration | before and after the 12 weeks intervention

CONTACTS AND LOCATIONS:
Overall Officials: Renger Witkamp, PhD, Principal Investigator — Wageningen University
Locations (1):
- Wageningen University, Division of Human Nutrition, Wageningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] de Bie TH, Witkamp RF, Balvers MG, Jongsma MA. Effects of gamma-aminobutyric acid supplementation on glucose control in adults with prediabetes: A double-blind, randomized, placebo-controlled trial. Am J Clin Nutr. 2023 Sep;118(3):708-719. doi: 10.1016/j.ajcnut.2023.07.017. Epub 2023 Jul 24. PMID 37495019
- [Derived] de Bie TH, Balvers MGJ, de Vos RCH, Witkamp RF, Jongsma MA. The influence of a tomato food matrix on the bioavailability and plasma kinetics of oral gamma-aminobutyric acid (GABA) and its precursor glutamate in healthy men. Food Funct. 2022 Aug 15;13(16):8399-8410. doi: 10.1039/d2fo01358d. PMID 35852458